CLINICAL TRIAL: NCT05528627
Title: Evaluation of the Efficacy of Pectoral Nerve (PECs) Blocks in Patients Undergoing Cardiac Implantable Electronic Device Insertion
Brief Title: PECs for Implantable Cardiac Electronic Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mustafa1
Record Dates: First submitted 2022-08-23; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Implantable Electronic Device; Nerve Block; Anesthesia; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pectoral Nerve (PECS) block (Other): Pectoral Nerve (PECs) block was performed at the surgical side 30 min before the procedure
  Interventions: Other: Pectoral Nerve (PECs) block

INTERVENTIONS:
Other: Pectoral Nerve (PECs) block — Pectoral Nerve (PECS) blocks were performed on the side of surgery, using the ultrasound-guided technique 30 min before the implantable cardiac electronic device (pacemaker, implantable cardioverter defibrillator) insertion procedure

SUMMARY:
The aim of this study is to evaluate the feasibility of the Pectoralis Nerve (PECS) block for CIED insertion.

DETAILED DESCRIPTION:
Implantable Cardiac Electronic Device (CIED) insertion can be performed under local anesthesia, regional anesthesia, or general anesthesia. Novel regional blocks may improve pain management for such patients and can shorten their length of stay in the hospital. At the study, the investigators aimd to evaluate the efficacy and feasibility of the PECS block for CIED insertion procedure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists grade II-IV patients
* in the age group of 18-80 years,
* Patients undergoing CIED insertion

Exclusion Criteria:

* pre-existing infection at the block site,
* coagulopathy,
* morbid obesity (Body mass index >35 kg m-2 ),
* allergy to local anaesthetics,
* decreased pulmonary reserve,
* psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
amount of intraoperative additional local anesthetic | 1 hour
  amount of intraoperative additional local anesthetic administered by the cardiologist during the CIED insertion procedure was recorded.
number of patients who requiring intraoperative additional local anesthetic | 1 hour
  Number of patients requiring intraoperative additional local anesthetic was recorded.

SECONDARY OUTCOMES:
Postoperative pain scores | 24 hours
  Postoperative pain scores were assessed by Visual Analogue Scale (VAS) scores from 0 (no pain) to 10 (maximum possible pain) for 24 hours postoperatively.
time to first postoperative analgesic requirement | 24 hours
  time to first postoperative analgesic requirement was recorded for 24 hours postoperatively
patient satisfaction | 24 hours
  Patient satisfaction was assessed by a 5-point Likert scale (ie, "1: very dissatisfied," "2: dissatisfied," "3: neutral," "4: satisfied," and "5: very satisfied") 24 hours after the procedure
cardiologist satisfaction | 24 hours
  Cardiologist satisfaction was assessed by a 5-point Likert scale (ie, "1: very dissatisfied," "2: dissatisfied," "3: neutral," "4: satisfied," and "5: very satisfied") 24 hours after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kilin, M.D., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)